CLINICAL TRIAL: NCT04271293
Title: anticOagulanti oRali in pazIenti fraGili Con gAstrostoMia endoscopIca Percutanea e fIbrillazione Atriale
Brief Title: Oral Anti-coagulants in Fragile Patients With Percutaneous Endoscopic Gastrostomy and Atrial Fibrillation (ORIGAMI) Pilot Study
Acronym: ORIGAMI
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, DAMARIO DOMENICO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2897
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PEG and oral anticoagulan treatment: Patients with PEG and indication for treatment with long-term oral anticoagulant therapy due to non valvular atrial fibrillation (FNAV), according to the current guidelines.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Edoxaban will be administered via PEG in patients who are eligible for the anticoagulant treatment according to the current guidelines.

SUMMARY:
Compelling evidences support the safety of direct oral anticoagulants (DOAC) compared to Vitamin K antagonists (VKA) in patients with non-valvular atrial fibrillation. The 2018 EHRA/ESC practical guide on the use of non-vitamin K antagonist oral anticoagulants stated that "data have shown that administration in a crushed form (e.g. via a nasogastric tube), does not alter the bioavailability for apixaban, rivaroxaban, and edoxaban". However, at the moment, there are no evidences supporting unequivocally the use of DOAC via PEG.

The purpose of this study is to evaluate the safety and efficacy of Edoxaban administered through PEG in patients with an indication of anticoagulation according to the current clinical practice.

DETAILED DESCRIPTION:
Several studies support the safety of direct oral anticoagulants (DOAC) compared to Vitamin K antagonists (VKA) in patients with non-valvular atrial fibrillation.

The 2018 EHRA/ESC practical guide on the use of non-vitamin K antagonist oral anticoagulants affirmed that "data have shown that administration in a crushed form (e.g. via a nasogastric tube), does not alter the bioavailability for apixaban, rivaroxaban, and edoxaban". However, at the moment, there are no evidences supporting unequivocally the use of DOAC via Percutaneous endoscopic gastrostomy (PEG).

PEG is a method developed throughout the early 1980s for patients who need long-term enteral nutrition due to neurodegenerative, neuromuscular and oncological diseases. This class of patients is expected to increase significantly in the next decade.

Several studies have proven the safety of DOAC compared to VKA even recommending to prefer DOAC over VKA wherever possible in the prevention of stroke and systemic embolism in adult patients with non-valvular atrial fibrillation. However, there is no evidence to support unequivocally the use of DOAC in patients fed PEG.

The purpose of this study is to evaluate the safety and efficacy of Edoxaban administered through PEG in patients with an indication of anticoagulation according to the current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PEG and indication for treatment with long-term oral anticoagulant therapy
* Patients with Atrial Fibrillation

Exclusion Criteria:

* Children under 18 years old.
* Life expectancy <30 days.
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Atrial Fibrillation. Patients with PEG and indication for treatment with long-term oral anticoagulant therapy according to the guidelines.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Cardio-embolic events | 1 month
  Description of the number of stroke, TIA and systemic embolism events symptomatic relapse of deep vein thrombosis/ pulmonary embolism in patients treated with Edoxaban via PEG.

SECONDARY OUTCOMES:
Bleeding events | 1 month
  any bleeding described according to the Bleeding Academic Research Consortium (BARC) scale.
  Type 0= No bleeding
  Type 1 = Bleeding that is not actionable and does not cause the patient to seek treatment.
  Type 2 = hemorrhage that "is actionable" and requires diagnostic studies, hospitalization, or treatment by a health care professional.
  Type 3a = bleeding plus hemoglobin drop of 3 to < 5 g/dl; transfusion with overt bleeding.
  Type 3b = bleeding plus hemoglobin drop < 5 g/dL; cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents.
  Type 3c = Confirmed Intracranial hemorrhage or intraocular bleed compromising vision
  Type 4 = CABG-related bleeding within 48 hours
  Type 5a = Probable fatal bleeding
  Type 5b = Definite fatal bleeding Type 0-2 will be conisdered minor bleedings. Type 3-5 will be considered major bleedings
Anti-factor Xa assay | within 1 month
  Description of the efficacy of the edoxaban by measuring th the anti-FXa activity.

CONTACTS AND LOCATIONS:
Overall Officials: Domenico D'Amario, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steffel J, Verhamme P, Potpara TS, Albaladejo P, Antz M, Desteghe L, Haeusler KG, Oldgren J, Reinecke H, Roldan-Schilling V, Rowell N, Sinnaeve P, Collins R, Camm AJ, Heidbuchel H; ESC Scientific Document Group. The 2018 European Heart Rhythm Association Practical Guide on the use of non-vitamin K antagonist oral anticoagulants in patients with atrial fibrillation. Eur Heart J. 2018 Apr 21;39(16):1330-1393. doi: 10.1093/eurheartj/ehy136. PMID 29562325
- [Background] Salmonson T, Dogne JM, Janssen H, Garcia Burgos J, Blake P. Non-vitamin-K oral anticoagulants and laboratory testing: now and in the future: Views from a workshop at the European Medicines Agency (EMA). Eur Heart J Cardiovasc Pharmacother. 2017 Jan;3(1):42-47. doi: 10.1093/ehjcvp/pvw032. Epub 2016 Dec 25. PMID 28025213
- [Background] Tripodi A, Ageno W, Ciaccio M, Legnani C, Lippi G, Manotti C, Marcucci R, Moia M, Morelli B, Poli D, Steffan A, Testa S. Position Paper on laboratory testing for patients on direct oral anticoagulants. A Consensus Document from the SISET, FCSA, SIBioC and SIPMeL. Blood Transfus. 2018 Sep;16(5):462-470. doi: 10.2450/2017.0124-17. Epub 2017 Sep 13. PMID 29106357
- [Background] Galli M, D'Amario D, Andreotti F, Porto I, Vergallo R, Sabatelli M, Lancellotti S, Meleo E, De Cristofaro R, Crea F. Sustained safe and effective anticoagulation using Edoxaban via percutaneous endoscopic gastrostomy. ESC Heart Fail. 2019 Aug;6(4):884-888. doi: 10.1002/ehf2.12434. Epub 2019 Jun 11. PMID 31184800
- [Derived] Cappannoli L, Laborante R, Galli M, Canonico F, Ciliberti G, Restivo A, Princi G, Arcudi A, Sabatelli M, De Cristofaro R, Crea F, D'Amario D. Feasibility, effectiveness, and safety of edoxaban administration through percutaneous endoscopic gastrostomy: 12-months follow up of the ORIGAMI study. Front Cardiovasc Med. 2022 Dec 22;9:1052053. doi: 10.3389/fcvm.2022.1052053. eCollection 2022. PMID 36620634
- [Derived] D'Amario D, Galli M, Canonico F, Restivo A, Arcudi A, Scacciavillani R, Cappannoli L, Riccioni ME, Annetta MG, Di Stefano G, Piccinni C, Vergallo R, Montone RA, Leone AM, Niccoli G, Sabatelli M, Antonelli M, Andreotti F, De Cristofaro R, Crea F. ORal anticoagulants In fraGile patients with percutAneous endoscopic gastrostoMy and atrIal fibrillation: the (ORIGAMI) study. J Cardiovasc Med (Hagerstown). 2021 Mar 1;22(3):175-179. doi: 10.2459/JCM.0000000000001142. PMID 33186237